CLINICAL TRIAL: NCT06666582
Title: Real-world Efficacy and Toxicity Data of the Combination of Paclitaxel and Ramucirumab Compared to Other Treatment Regimens in Patients With Advanced Gastric Cancer
Brief Title: Real-world Data of Paclitaxel and Ramucirumab Compared to Other Treatment Regimens in Advanced Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: RE721
Record Dates: First submitted 2024-04-09; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer Stage IV; Second-line Treatment; Ramucirumab Paclitaxel
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Ramucirumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who received paclitaxel - ramucirumab as second-line treatment: Patients with unresectable or metastatic, locally advanced adenocarcinoma of the stomach, gastroesophageal junction, or distal esophagus who had been treated at Departments of Medical Oncology affiliated with the Hellenic Cooperative Oncology Group (HeCOG). All patients had received second-line treatment for advanced disease with paclitaxel and ramucirumab, for at least two months.
  Interventions: Drug: Paclitaxel and ramucirumab
- Patients who received other regimens as second-line treatment: patients with unresectable or metastatic, locally advanced adenocarcinoma of the stomach, gastroesophageal junction, or distal esophagus who had been treated at Departments of Medical Oncology affiliated with the Hellenic Cooperative Oncology Group (HeCOG). All patients had received second-line treatment for advanced disease based on international/national guidelines, except from paclitaxel and ramucirumab. All other regimens, combinations of drugs as well as monotherapy, were accepted. Patients were included in the analysis if they have received at least two months of second-line treatment.
  Interventions: Drug: Paclitaxel and ramucirumab

INTERVENTIONS:
Drug: Paclitaxel and ramucirumab — Second-line treatment with paclitaxel/ramucirumab vs other regimens

SUMMARY:
Our aim was to evaluate whether second-line treatment with paclitaxel and ramucirumab was associated with improved clinical outcomes compared to other available therapies. This study involved real-world data collection, focusing on the safety and efficacy of therapeutic combinations, administered to patients with pretreated advanced gastric cancer in the Oncology Departments affiliated with the Hellenic Cooperative Oncology Group (HeCOG).

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic, locally advanced adenocarcinoma of the stomach, gastroesophageal junction, or distal esophagus
* Treated at Departments of Medical Oncology affiliated with the Hellenic Cooperative Oncology Group (HeCOG)
* Second-line treatment for advanced disease
* Treatment for at least two months of second-line treatment.

Exclusion Criteria:

* Lack of informed consent in case the patient was alive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients with unresectable or metastatic, locally advanced adenocarcinoma of the stomach, gastroesophageal junction, or distal esophagus who had been treated at Departments of Medical Oncology affiliated with the Hellenic Cooperative Oncology Group (HeCOG). All patients had received second-line treatment for advanced disease based on international/national guidelines. All regimens, combinations of drugs as well as monotherapy, were accepted. Patients were included in the analysis if they have received at least two months of second-line treatment. Patient clinicopathological characteristics and outcome data were retrospectively recorded from patient medical records. Toxicity data were retrospectively recorded from the clinicians' documentations of patient-reported symptoms and laboratory results during scheduled clinical visits or patient hospitalizations.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From the initiation of second-line treatment to the date of discontinuation (due to any reason), first documented progression, death from any cause or last contact, through study completion, up to 2 years
  The primary endpoint of interest was the assessment of progression-free survival (PFS1), defined as the time interval from the initiation of second-line treatment to the date of discontinuation (due to any reason), first documented progression, death from any cause or last contact, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | From the date of disease progression to the date of death from any cause or last contact, through study completion, up to 2 years.
  overall survival (OS), defined as the time interval from the date of disease progression to the date of death from any cause or last contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Oncology Cooperative Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Could share anonymized clinical data upon request, after approval by our institutions